CLINICAL TRIAL: NCT01721044
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study Evaluating the Efficacy and Safety of Baricitinib (LY3009104) in Patients With Moderately to Severely Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Tumor Necrosis Factor Inhibitors
Brief Title: A Moderate to Severe Rheumatoid Arthritis Study
Acronym: RA-BEACON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14058; I4V-MC-JADW (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-11-01; First posted 2012-11-02 (Estimated); Results first posted 2018-01-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo administered orally once daily through Week 24. Starting at Week 16, participants who are nonresponders will be rescued with baricitinib 4 milligram (mg) orally once daily through Week 24.
  Participants will continue to take background conventional disease-modifying antirheumatic drug (cDMARD) therapy throughout study.
  Interventions: Drug: Placebo; Drug: cDMARD
- Baricitinib 2 mg (Experimental): Baricitinib 2 mg administered orally once daily through Week 24. Starting at Week 16, participants who are nonresponders will be rescued with baricitinib 4 mg orally once daily through Week 24.
  Participants will continue to take background cDMARD therapy throughout study.
  Interventions: Drug: Baricitinib; Drug: cDMARD
- Baricitinib 4 mg (Experimental): Baricitinib 4 mg administered orally once daily through Week 24. Starting at Week 16, participants who are nonresponders will be rescued with baricitinib 4 mg orally once daily through Week 24.
  Participants will continue to take background cDMARD therapy throughout study.
  Interventions: Drug: Baricitinib; Drug: cDMARD

INTERVENTIONS:
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: Baricitinib — Administered orally
  Other Names: LY 3009104; INCB 028050
  Arms: Baricitinib 2 mg; Baricitinib 4 mg
Drug: cDMARD — Participants will continue to take background cDMARD therapy throughout study.

SUMMARY:
The purpose of this study is to determine whether baricitinib 4 milligram (mg) once daily is superior to placebo in the treatment of participants with moderately to severely active Rheumatoid Arthritis (RA) who have had an inadequate response to a tumor necrosis factor (TNF) inhibitor, despite ongoing treatment with conventional disease-modifying antirheumatic drugs (cDMARDs).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of adult-onset Rheumatoid Arthritis (RA) as defined by the American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR) 2010 Criteria for the Classification of RA
* Have moderately to severely active RA defined as the presence of at least 6/68 tender joints and at least 6/66 swollen joints
* Have a C-reactive protein (CRP) or high-sensitivity C-reactive protein (hsCRP) measurement ≥ (greater than or equal to) 1 times the upper limit of normal (ULN)
* Have been treated at approved doses with at least 1 biologic tumor necrosis factor (TNF)- alpha inhibitor for at least 3 months and either:

  * experienced insufficient efficacy or loss of efficacy
  * experienced intolerance of such treatment
* Have had regular use of at least 1 conventional disease-modifying antirheumatic drugs (cDMARD) for at least the 12 weeks prior to study entry with a continuous, nonchanging dose for at least 8 weeks prior to study entry

Exclusion Criteria:

* Have received a biologic treatment for RA within 28 days of planned randomization; have received rituximab within 6 months of planned randomization
* Are currently receiving corticosteroids at doses > (greater than) 10 mg per day of prednisone (or equivalent) or have been receiving an unstable dosing regimen of corticosteroids within 2 weeks of study entry or within 6 weeks of planned randomization
* Have started treatment with non-steroidal anti-inflammatory drugs (NSAIDs) or have been receiving an unstable dosing regimen of NSAIDs within 2 weeks of study entry or within 6 weeks of planned randomization
* Are currently receiving concomitant treatment with methotrexate (MTX), hydroxychloroquine, and sulfasalazine or combination of any 3 cDMARDs
* Have received any parenteral corticosteroid administered by intramuscular or intravenous (IV) injection within 2 weeks prior to study entry or within 6 weeks prior to planned randomization or are anticipated to require parenteral injection of corticosteroids during the study
* Have had 3 or more joints injected with intraarticular corticosteroids or hyaluronic acid within 2 weeks prior to study entry or within 6 weeks prior to planned randomization
* Have active fibromyalgia that, in the investigator's opinion, would make it difficult to appropriately assess RA activity for the purposes of this study
* Have a diagnosis of any systemic inflammatory condition other than RA, such as, but not limited to juvenile chronic arthritis, spondyloarthropathy, Crohn's disease, ulcerative colitis, psoriatic arthritis, active vasculitis or gout (participants with secondary Sjogren's syndrome are not excluded.)
* Have a diagnosis of Felty's syndrome
* Have had any major surgery within 8 weeks of study entry or will require major surgery during the study that, in the opinion of the investigator in consultation with Lilly or its designee, would pose an unacceptable risk to the participant
* Have experienced any of the following within 12 weeks of study entry: myocardial infarction, unstable ischemic heart disease, stroke, or have New York Heart Association stage IV heart failure
* Have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute a risk when taking investigational product or could interfere with the interpretation of data
* Are largely or wholly incapacitated permitting little or no self care, such as, being bedridden or confined to a wheelchair
* Have an estimated glomerular filtration rate (eGFR) based on the most recent available serum creatinine using the Modification of Diet in Renal Disease (MDRD) method of < (less than) 40 milliliter per minute per 1.73 m^2 (mL/min/1.73 m^2)
* Have a history of chronic liver disease with the most recent available aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 times the ULN or the most recent available total bilirubin ≥1.5 times the ULN
* Have a history of, lymphoproliferative disease; or have signs or symptoms suggestive of possible lymphoproliferative disease, including lymphadenopathy or splenomegaly; or have active primary or recurrent malignant disease; or have been in remission from clinically significant malignancy for <5 years
* Have been exposed to a live vaccine within 12 weeks prior to planned randomization or are expected to need/receive a live vaccine during the course of the study (with the exception of herpes zoster vaccination)
* Have a current or recent clinically serious viral, bacterial, fungal, or parasitic infection
* Have had symptomatic herpes zoster infection within 12 weeks prior to study entry
* Have a history of disseminated/complicated herpes zoster (eg, multidermatomal involvement, ophthalmic zoster, central nervous system involvement, postherpetic neuralgia)
* Are immunocompromised and, in the opinion of the investigator, are at an unacceptable risk for participating in the study
* Have a history of active hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)
* Have screening laboratory test values, including thyroid-stimulating hormone (TSH), outside the reference range for the population or investigative site that, in the opinion of the investigator, pose an unacceptable risk for the participant's participation in the study
* Have screening electrocardiogram (ECG) abnormalities that, in the opinion of the investigator or the sponsor, are clinically significant and indicate an unacceptable risk for the participant's participation in the study (e.g. Fridericia's corrected QT interval >500 millisecond [msec])
* Have symptomatic herpes simplex at the time of study enrollment
* Have evidence of active or latent tuberculosis (TB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (103):
- United States (32):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palo Alto, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Upland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danbury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trumbull, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lewes, Delaware
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boynton Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tamarac, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boise, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lansing, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freehold, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hartsdale, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tulsa, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethlehem, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wyomissing, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Myrtle Beach, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nassau Bay, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Webster, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chesapeake, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kennewick, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Franklin, Wisconsin
- Argentina (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kogarah, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maroochydore, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fitzroy, Victoria
- Austria (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mons
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario, Canada
- Denmark (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frederiksberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glostrup Municipality
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odense
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orléans
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tours
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Würzburg
- Greece (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heraklion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kifissia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Larissa
- Israel (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ashkelon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beer Yaakov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerusalem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kfar Saba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petah Tikva
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Aviv
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- Japan (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Japan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- Mexico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ubbergen, Netherlands
- Poland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nadarzyn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Puerto Rico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caguas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santurce
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santander
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villajoyosa
- Switzerland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fribourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lausanne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zurich
- Turkey (Türkiye) (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edirne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gaziantep
- United Kingdom (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Shields, Tyneside
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bradford, West Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Taylor PC, Takeuchi T, Burmester GR, Durez P, Smolen JS, Deberdt W, Issa M, Terres JR, Bello N, Winthrop KL. Safety of baricitinib for the treatment of rheumatoid arthritis over a median of 4.6 and up to 9.3 years of treatment: final results from long-term extension study and integrated database. Ann Rheum Dis. 2022 Mar;81(3):335-343. doi: 10.1136/annrheumdis-2021-221276. Epub 2021 Oct 27. PMID 34706874
- [Derived] Wells AF, Jia B, Xie L, Valenzuela GJ, Keystone EC, Li Z, Quebe AK, Griffing K, Otawa S, Haraoui B. Efficacy of Long-Term Treatment with Once-Daily Baricitinib 2 mg in Patients with Active Rheumatoid Arthritis: Post Hoc Analysis of Two 24-Week, Phase III, Randomized, Controlled Studies and One Long-Term Extension Study. Rheumatol Ther. 2021 Jun;8(2):987-1001. doi: 10.1007/s40744-021-00317-9. Epub 2021 May 24. PMID 34028703
- [Derived] Emery P, Tanaka Y, Cardillo T, Schlichting D, Rooney T, Beattie S, Helt C, Smolen JS. Temporary interruption of baricitinib: characterization of interruptions and effect on clinical outcomes in patients with rheumatoid arthritis. Arthritis Res Ther. 2020 May 15;22(1):115. doi: 10.1186/s13075-020-02199-8. PMID 32414425
- [Derived] Smolen JS, Genovese MC, Takeuchi T, Hyslop DL, Macias WL, Rooney T, Chen L, Dickson CL, Riddle Camp J, Cardillo TE, Ishii T, Winthrop KL. Safety Profile of Baricitinib in Patients with Active Rheumatoid Arthritis with over 2 Years Median Time in Treatment. J Rheumatol. 2019 Jan;46(1):7-18. doi: 10.3899/jrheum.171361. Epub 2018 Sep 15. PMID 30219772
- [Derived] Tanaka Y, McInnes IB, Taylor PC, Byers NL, Chen L, de Bono S, Issa M, Macias WL, Rogai V, Rooney TP, Schlichting DE, Zuckerman SH, Emery P. Characterization and Changes of Lymphocyte Subsets in Baricitinib-Treated Patients With Rheumatoid Arthritis: An Integrated Analysis. Arthritis Rheumatol. 2018 Dec;70(12):1923-1932. doi: 10.1002/art.40680. Epub 2018 Oct 22. PMID 30058112
- [Derived] Taylor PC, Kremer JM, Emery P, Zuckerman SH, Ruotolo G, Zhong J, Chen L, Witt S, Saifan C, Kurzawa M, Otvos JD, Connelly MA, Macias WL, Schlichting DE, Rooney TP, de Bono S, McInnes IB. Lipid profile and effect of statin treatment in pooled phase II and phase III baricitinib studies. Ann Rheum Dis. 2018 Jul;77(7):988-995. doi: 10.1136/annrheumdis-2017-212461. Epub 2018 Feb 20. PMID 29463520
- [Derived] Genovese MC, Kremer JM, Kartman CE, Schlichting DE, Xie L, Carmack T, Pantojas C, Sanchez Burson J, Tony HP, Macias WL, Rooney TP, Smolen JS. Response to baricitinib based on prior biologic use in patients with refractory rheumatoid arthritis. Rheumatology (Oxford). 2018 May 1;57(5):900-908. doi: 10.1093/rheumatology/kex489. PMID 29415145
- [Derived] Smolen JS, Kremer JM, Gaich CL, DeLozier AM, Schlichting DE, Xie L, Stoykov I, Rooney T, Bird P, Sanchez Burson JM, Genovese MC, Combe B. Patient-reported outcomes from a randomised phase III study of baricitinib in patients with rheumatoid arthritis and an inadequate response to biological agents (RA-BEACON). Ann Rheum Dis. 2017 Apr;76(4):694-700. doi: 10.1136/annrheumdis-2016-209821. Epub 2016 Oct 31. PMID 27799159
- [Derived] Genovese MC, Kremer J, Zamani O, Ludivico C, Krogulec M, Xie L, Beattie SD, Koch AE, Cardillo TE, Rooney TP, Macias WL, de Bono S, Schlichting DE, Smolen JS. Baricitinib in Patients with Refractory Rheumatoid Arthritis. N Engl J Med. 2016 Mar 31;374(13):1243-52. doi: 10.1056/NEJMoa1507247. PMID 27028914

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who did not adequately respond (nonresponders) to study drug were eligible for rescue treatment with baricitinib 4 mg beginning at Week 16. Nonresponders were defined as lack of improvement of at least 20% in both tender joint count and swollen joint count at both Weeks 14 and 16 compared to baseline.
Groups:
- Placebo: Placebo administered orally (PO) once daily (QD) through Week 24. Participants continued to take background conventional disease-modifying antirheumatic drug (cDMARD) therapy throughout study.
- Baricitinib 2 mg: Baricitinib 2 milligram (mg) administered PO QD through Week 24. Participants continued to take background cDMARD therapy throughout study.
- Baricitinib 4 mg: Baricitinib 4 mg administered PO QD through Week 24. Participants continued to take background cDMARD therapy throughout study.
Period: Treatment Period
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Started | 176 | 174 (Randomized to 4mg (N=11) but received 2mg due to moderate renal impairment were included in 4mg arm) | 177
Rescue Week 16-24 | 56 | 38 | 33
Completed | 144 | 157 | 158
Not Completed | 32 | 17 | 19
Not completed — Adverse Event | 7 | 7 | 10
Not completed — Death | 0 | 0 | 1
Not completed — Lack of Efficacy | 16 | 4 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 6 | 1
Period: Follow Up
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Started | 19 (Participants from treatment who entered the post-treatment follow-up period.) | 9 (Participants from treatment who entered the post-treatment follow-up period.) | 20 (Participants from treatment and rescue who entered the post-treatment follow-up period.)
Completed | 19 | 9 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) population includes all randomized participants who received at least 1 dose of the study drug.
Groups:
- Placebo: Placebo administered PO QD through Week 24. Participants continued to take background cDMARD therapy throughout study.
- Baricitinib 2 mg: Baricitinib 2 mg administered PO QD through Week 24. Participants continued to take background cDMARD therapy throughout study.
- Total: Total of all reporting groups
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg | Total
Number analyzed (Participants) | 176 | 174 | 177 | 527
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.0 (10.7) | 55.1 (11.1) | 55.9 (11.3) | 55.7 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 137 | 149 | 431
  Male | 31 | 37 | 28 | 96
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 12 | 11 | 32
  Asian | 11 | 9 | 12 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 9 | 7 | 24
  White | 147 | 144 | 144 | 435
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 9 | 5 | 7 | 21
  Australia | 8 | 9 | 4 | 21
  Austria | 5 | 3 | 8 | 16
  Belgium | 1 | 1 | 1 | 3
  Canada | 1 | 4 | 3 | 8
  Denmark | 2 | 3 | 1 | 6
  France | 7 | 10 | 7 | 24
  Germany | 8 | 5 | 6 | 19
  Greece | 4 | 3 | 2 | 9
  Israel | 9 | 8 | 13 | 30
  Italy | 2 | 3 | 3 | 8
  Japan | 6 | 6 | 8 | 20
  Mexico | 9 | 12 | 10 | 31
  Netherlands | 0 | 1 | 1 | 2
  Poland | 10 | 13 | 9 | 32
  South Korea | 4 | 3 | 3 | 10
  Spain | 10 | 7 | 10 | 27
  Switzerland | 1 | 2 | 4 | 7
  Turkey | 1 | 1 | 1 | 3
  United Kingdom | 2 | 1 | 1 | 4
  United States | 77 | 74 | 75 | 226
Duration of Rheumatoid Arthritis [Mean (Standard Deviation); unit: Years] — Time from Symptom Onset of Rheumatoid Arthritis
  Years | 14.0 (9.6) | 13.7 (8.0) | 14.3 (9.4) | 14.0 (9.0)
Tender Joint Count of 68 Evaluable Joints [Mean (Standard Deviation); unit: Number of Joints] — Population: Tender joint count based on 68 joints.
  Number of Joints
    number analyzed (Participants) | 174 | 174 | 177 | 525
    (all) | 28.3 (16.4) | 31.0 (16.3) | 28.1 (15.6) | 29.1 (16.1)
Swollen Joint Count of 66 Evaluable Joints [Mean (Standard Deviation); unit: Number of Joints] — Population: Swollen joint count based on 66 joints.
  Number of Joints
    number analyzed (Participants) | 174 | 174 | 177 | 525
    (all) | 17.2 (10.8) | 18.6 (12.3) | 16.3 (8.9) | 17.4 (10.8)
High Sensitivity C-Reactive Protein (hsCRP) [Mean (Standard Deviation); unit: milligrams/liter (mg/L)] | 20.64 (25.26) | 19.87 (22.48) | 19.76 (24.84) | 20.09 (24.19)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response - Placebo Versus Baricitinib 4 mg
Description: ACR20 Responder Index is a composite of clinical, laboratory, and functional measures in rheumatoid arthritis. ACR20 Responder is a participant who has at least 20% improvement in both tender and swollen joint counts and in at least 3 of the following 5 criteria: Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity using visual analog scale (VAS), Health Assessment Questionnaire - Disability Index (HAQ-DI), pain due to arthritis, and high-sensitivity C-reactive protein (hsCRP). Participants with missing responses and participants who discontinue study or drug or are rescued before analysis timepoint are deemed non-responders.
Time Frame: Week 12
Population: Modified Intent-to-Treat (mITT) population includes all randomized participants who received at least 1 dose of the study drug. Participants will be analyzed according to the study drug to which they were randomized. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using non-responder imputation (NRI).
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Baricitinib 4 mg
Number analyzed (Participants) | 176 | 177
Percentage of Participants | 27.3 | 55.4
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; Test type: Superiority or Other; p = 0.001, Regression, Logistic; If logistic regression sample size requirements are not met, the p-value from Fisher's exact test is used instead

2. Secondary Outcome: Change From Baseline in HAQ-DI Score - Placebo Versus Baricitinib 4 mg
Description: The HAQ-DI questionnaire assesses the participant's self-perception on the degree of difficulty [0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do)] when dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and performing other daily activities. Scores for each functional area were averaged to calculate the HAQ-DI score, which ranged from 0 (no disability) to 3 (worst disability). A decrease in HAQ-DI score indicated an improvement in the participant's condition.
Time Frame: Baseline, Week 12
Population: mITT population includes all randomized participants who received at least 1 dose of the study drug. Participants were analyzed according to the study drug to which they were randomized. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using modified baseline observation carried forward (mBOCF).
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Baricitinib 4 mg
Number analyzed (Participants) | 176 | 177
Units on a Scale | -0.20 (0.50) | -0.42 (0.49)
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; Test type: Superiority or Other; p = 0.001, ANCOVA

3. Secondary Outcome: Change From Baseline in the Disease Activity Score Based on a 28-Joint Count (DAS-28) High Sensitivity C-Reactive Protein (hsCRP) - Placebo Versus Baricitinib 4 mg
Description: DAS-28 consisted of composite score of following variables: tender joint count (TJC28), swollen joint count (SJC28), high sensitivity C-reactive protein (hsCRP) (milligrams per liter), and Patient's Global Assessment of Disease Activity. DAS28 was calculated using following formula: DAS28-hsCRP=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(CRP+1)+0.014*Patient's Global VAS+0.96. Total scores ranged from 1.0-9.4, where lower scores indicated less disease activity.
Time Frame: Baseline, Week 12
Population: mITT population includes all randomized participants who received at least 1 dose of the study drug. Participants were analyzed according to the study drug to which they were randomized. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using mBOCF.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Baricitinib 4 mg
Number analyzed (Participants) | 174 | 177
Units on a Scale | -0.85 (1.19) | -1.81 (1.43)
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; Test type: Superiority or Other; p = 0.001, ANCOVA

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Remission - Simplified Disease Activity Index (SDAI) ≤3.3 - Placebo Versus Baricitinib 4 mg
Description: The ACR/EULAR definitions of rheumatoid arthritis (RA) remission includes an index-based definition. The index-based definition of remission occurs with a SDAI score ≤3.3. The SDAI is a tool for measurement of disease activity in RA that integrates TJC28 (0 to 28), SJC28 (0 to 28), acute phase response using C-reactive protein (0.1 to 10.0 mg/dL), Patient's Global Assessment of Disease Activity using VAS (0 to 10.0 cm), and Physician's Global Assessment of Disease Activity using VAS (0 to 10.0 cm). Lower scores indicated less disease activity.
Time Frame: Week 12
Population: mITT population includes all randomized participants who received at least 1 dose of the study drug. Participants were analyzed according to the study drug to which they were randomized or assigned per protocol. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using NRI.
Measure: Number; unit: Percent of Participants
Arm/Group | Placebo | Baricitinib 4 mg
Number analyzed (Participants) | 176 | 177
Percent of Participants | 1.7 | 5.1
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; Test type: Superiority or Other; p = 0.140, Regression, Logistic; If logistic regression sample size requirements are not met, the p-value from Fisher's exact test is used instead

5. Secondary Outcome: Percentage of Participants Achieving ACR20 Response - Placebo Versus Baricitinib 2 mg
Description: ACR20 Responder Index is a composite of clinical, laboratory, and functional measures in rheumatoid arthritis. ACR20 Responder is a participant who has at least 20% improvement in both tender and swollen joint counts and in at least 3 of the following 5 criteria: Physician's Global Assessment of Disease Activity using VAS, Patient's Global Assessment of Disease Activity using VAS, HAQ-DI, pain due to arthritis, and hsCRP. Participants with missing responses and participants who discontinue study or drug or are rescued before analysis time point are deemed non-responders.
Time Frame: Week 12
Population: Modified Intent-to-Treat (mITT) population includes all randomized participants who received at least 1 dose of the study drug. Participants will be analyzed according to the study drug to which they were randomized. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using NRI.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Baricitinib 2 mg
Number analyzed (Participants) | 176 | 174
Percentage of Participants | 27.3 | 48.9
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 2 mg; Test type: Superiority or Other; p = 0.001, Regression, Logistic; If logistic regression sample size requirements are not met, the p-value from Fisher's exact test is used instead

6. Secondary Outcome: Change From Baseline in HAQ-DI Score - Placebo Versus Baricitinib 2 mg
Description: The HAQ-DI questionnaire assesses the participant's self-perception on the degree of difficulty [0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do)] when dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and performing other daily activities. Scores for each functional area were averaged to calculate the HAQ-DI score. Total scores ranged from 0 (no disability) to 3 (worst disability). A decrease in HAQ-DI score indicated an improvement in the participant's condition.
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Baricitinib 2 mg
Number analyzed (Participants) | 176 | 174
Units on a Scale | -0.20 (0.50) | -0.38 (0.51)
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 2 mg; Test type: Superiority or Other; p = 0.001, ANCOVA

7. Secondary Outcome: Change From Baseline in the DAS28 - hsCRP - Placebo Versus Baricitinib 2 mg
Description: DAS28 consisted of composite score of following variables: TJC28, SJC28, hsCRP (mg/mL), and Patient's Global Assessment of Disease Activity. DAS28 was calculated using following formula: DAS28-CRP=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(CRP+1)+0.014*Patient's Global VAS+0.96. Total scores ranged from 1.0-9.4, where lower scores indicated less disease activity.
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Baricitinib 2 mg
Number analyzed (Participants) | 176 | 174
Units on a Scale | -0.85 (1.19) | -1.53 (1.34)
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 2 mg; Test type: Superiority or Other; p = 0.001, ANCOVA

8. Secondary Outcome: Percentage of Participants Achieving ACR/EULAR Remission - SDAI ≤3.3 - Placebo Versus Baricitinib 2 mg
Description: as for outcome 4
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: Percent of Participants
Arm/Group | Placebo | Baricitinib 2 mg
Number analyzed (Participants) | 176 | 174
Percent of Participants | 1.7 | 2.3
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 2 mg; Test type: Superiority or Other; p = 0.723, Regression, Logistic; If logistic regression sample size requirements are not met, the p-value from Fisher's exact test is used instead

9. Secondary Outcome: Percentage of Participants Achieving ACR20 Response
Description: as for outcome 5
Time Frame: Week 24
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 176 | 174 | 177
Percentage of Participants | 27.3 | 44.8 | 46.3
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; Test type: Superiority or Other; p = 0.001, Regression, Logistic — a priori p-value significance threshold: 2-sided <=0.05; If logistic regression sample size requirements are not met, the p-value from Fisher's exact test is used instead
Statistical Analysis 2: Comparison: Placebo vs Baricitinib 2 mg; Test type: Superiority or Other; p = 0.001, Regression, Logistic — a priori p-value significance threshold: 2-sided <=0.05; If logistic regression sample size requirements are not met, the p-value from Fisher's exact test is used instead

10. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response
Description: ACR50 Responder Index is a composite of clinical, laboratory, and functional measures in RA. ACR50 Responder is a participant who has at least 50% improvement in both tender and swollen joint counts and in at least 3 of the following 5 criteria: Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity, HAQ-DI, pain due to arthritis, and hsCRP. Participants with missing responses and participants who discontinue study or drug or are rescued before analysis time point are deemed non-responders.
Time Frame: Week 12 and Week 24
Population: mITT population includes all randomized participants who received at least 1 dose of the study drug. Participants were analyzed according to the study drug to which they were randomized. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using NRI.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 176 | 174 | 177
Percentage of Participants
  Week 12 | 8.0 | 20.1 | 28.2
  Week 24 | 13.1 | 23.0 | 29.4
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; Week 12; Test type: Superiority or Other; p = 0.001, Regression, Logistic — a priori p-value significance threshold: 2-sided ≤0.05; If logistic regression sample size requirements are not met, the p-value from Fisher's exact test is used instead
Statistical Analysis 2: Comparison: Placebo vs Baricitinib 2 mg; Week 12; Test type: Superiority or Other; p = 0.002, Regression, Logistic — a priori p-value significance threshold: 2-sided ≤0.05; If logistic regression sample size requirements are not met, the p-value from Fisher's exact test is used instead
Statistical Analysis 3: Comparison: Placebo vs Baricitinib 4 mg; Week 24; Test type: Superiority or Other; p = 0.001, Regression, Logistic — a priori p-value significance threshold: 2-sided ≤0.05; If logistic regression sample size requirements are not met, the p-value from Fisher's exact test is used instead
Statistical Analysis 4: Comparison: Placebo vs Baricitinib 2 mg; Week 24; Test type: Superiority or Other; p = 0.015, Regression, Logistic — a priori p-value significance threshold: 2-sided ≤0.05; If logistic regression sample size requirements are not met, the p-value from Fisher's exact test is used instead

11. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response
Description: ACR70 Responder Index is a composite of clinical, laboratory, and functional measures in RA. ACR70 Responder is a participant who has at least 70% improvement in both tender and swollen joint counts and in at least 3 of the following 5 criteria: Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity, HAQ-DI, pain due to arthritis, and hsCRP. Participants with missing responses and participants who discontinue study or drug or are rescued before analysis time point are deemed non-responders.
Time Frame: Week 12 and Week 24
Population: as for outcome 10
Measure: Number; unit: Percentage of Participants
Groups:
- Placebo: Placebo administered PO QD through Week 24. Participants will continue to take background cDMARD therapy throughout study.
- Baricitinib 2 mg: Baricitinib 2 mg administered PO QD through Week 24. Participants will continue to take background cDMARD therapy throughout study.
- Baricitinib 4 mg: Baricitinib 4 mg administered PO QD through Week 24. Participants will continue to take background cDMARD therapy throughout study.
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 176 | 174 | 177
Percentage of Participants
  Week 12 | 2.3 | 12.6 | 11.3
  Week 24 | 3.4 | 13.2 | 16.9
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; Week 12; Test type: Superiority or Other; p = 0.002, Regression, Logistic — a priori p-value significance threshold: 2-sided ≤0.05; If logistic regression sample size requirements are not met, the p-value from Fisher's exact test is used instead
Statistical Analysis 2: Comparison: Placebo vs Baricitinib 2 mg; Week 12; Test type: Superiority or Other; p = 0.001, Regression, Logistic — a priori p-value significance threshold: 2-sided ≤0.05; If logistic regression sample size requirements are not met, the p-value from Fisher's exact test is used instead
Statistical Analysis 3: Comparison: Placebo vs Baricitinib 4 mg; Week 24; Test type: Superiority or Other; p = 0.001, Regression, Logistic — a priori p-value significance threshold: 2-sided ≤0.05; If logistic regression sample size requirements are not met, the p-value from Fisher's exact test is used instead
Statistical Analysis 4: Comparison: Placebo vs Baricitinib 2 mg; Week 24; Test type: Superiority or Other; p = 0.001, Regression, Logistic — a priori p-value significance threshold: 2-sided ≤0.05; If logistic regression sample size requirements are not met, the p-value from Fisher's exact test is used instead

12. Secondary Outcome: Change From Baseline in DAS28 - Erythrocyte Sedimentation Rate (ESR)
Description: DAS28 consisted of composite score of following variables: tender joint count (TJC28), swollen joint count (SJC28), ESR (millimeters per hour), and Patient's Global Assessment of Disease Activity. DAS28 was calculated using following formula: DAS28-ESR=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.70*natural log(ESR)+0.014*Patient's Global VAS. Total scores ranged from 1.0-9.4, where lower scores indicated less disease activity.
Time Frame: Baseline, Week 12
Population: mITT population includes all randomized participants who received at least 1 dose of the study drug. Participants were analyzed according to the study drug to which they were randomized. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using modified last observation carried forward (mLOCF).
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 168 | 169 | 173
Units on a Scale | -0.92 (1.21) | -1.52 (1.37) | -1.80 (1.44)
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; Test type: Superiority or Other; p = 0.001, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05
Statistical Analysis 2: Comparison: Placebo vs Baricitinib 2 mg; Test type: Superiority or Other; p = 0.001, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05

13. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index Score
Description: The CDAI is a tool for measurement of disease activity in RA that does not require a laboratory component and was scored by the investigative site. It integrates TJC28 (scored 0-28 with higher scores indicating higher disease activity), SJC28 (scored 0-28 with higher scores indicating higher disease activity), Patient's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity), and Physician's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity). The CDAI is calculated by summing the values of the 4 components. CDAI scores range from 0 to 76; lower scores indicated lower disease activity. A negative change from baseline indicates improvement in condition.
Time Frame: Baseline, Week 24
Population: mITT population includes all randomized participants who received at least 1 dose of the study drug. Participants were analyzed according to the study drug to which they were randomized. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using mLOCF.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 170 | 169 | 171
Units on a Scale | -12.19 (16.96) | -17.17 (16.96) | -20.30 (16.29)
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; Test type: Superiority or Other; p = 0.001, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05
Statistical Analysis 2: Comparison: Placebo vs Baricitinib 2 mg; Test type: Superiority or Other; p = 0.009, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05

14. Secondary Outcome: Change From Baseline in Measures of SDAI Score
Description: The SDAI is a tool for measurement of disease activity in RA that integrates TJC28, SJC28, acute phase response using C-reactive protein (milligrams per liter), Patient's Global Assessment of Disease Activity using visual analog scale (cm), and Physician's Global Assessment of Disease Activity using visual analog scale (cm). The SDAI is calculated by summing the values of the 5 components. Lower scores indicated less disease activity.
  The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst). A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 170 | 169 | 171
Units on a Scale | -12.07 (17.50) | -17.80 (17.50) | -21.26 (17.01)
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; Test type: Superiority or Other; p = 0.001, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05
Statistical Analysis 2: Comparison: Placebo vs Baricitinib 2 mg; Test type: Superiority or Other; p = 0.003, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05

15. Secondary Outcome: Percentage of Participants Achieving ACR/EULAR Remission - Boolean Remission
Description: The ACR/EULAR definitions of RA remission includes a Boolean-based definition. The Boolean-based definition of remission occurs when all 4 of the following criteria are met at the same visit: TJC28 ≤1, SJC28 ≤1, acute phase response using C-reactive protein (milligrams per deciliter) ≤1, Patient's Global Assessment of Disease Activity using VAS (cm) ≤1.
Time Frame: Week 24
Population: as for outcome 10
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 176 | 174 | 177
Percentage of Participants | 1.1 | 4.0 | 6.8
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; Test type: Superiority or Other; p = 0.012, Regression, Logistic — a priori p-value significance threshold: 2-sided ≤0.05; If logistic regression sample size requirements are not met, the p-value from Fisher's exact test is used instead
Statistical Analysis 2: Comparison: Placebo vs Baricitinib 2 mg; Test type: Superiority or Other; p = 0.104, Regression, Logistic — a priori p-value significance threshold: 2-sided ≤0.05; If logistic regression sample size requirements are not met, the p-value from Fisher's exact test is used instead

16. Secondary Outcome: Change From Baseline in Duration of Participant Reported Outcome - Morning Joint Stiffness
Description: Participants reported the duration of their morning joint stiffness (MJS) in hours and minutes. The participants were asked about their duration of morning joint stiffness on the day prior to the study visit to capture actual symptoms, since the participant may have had an atypical morning routine on that day. If morning joint stiffness duration was longer than 12 hours (720 minutes), it was truncated to 720 minutes for statistical presentations and analyses. A decrease in duration of morning joint stiffness indicated an improvement in the participant's condition.
Time Frame: Baseline, Week 24
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 172 | 172 | 175
Minutes | -8.0 [-15.0 to 0.0] | -25.5 [-40.0 to -15.0] | -27.0 [-40.0 to -15.0]
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney) — a priori p-value significance threshold: 2-sided ≤0.05
Statistical Analysis 2: Comparison: Placebo vs Baricitinib 2 mg; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney) — a priori p-value significance threshold: 2-sided ≤0.05

17. Secondary Outcome: Change From Baseline in Worst Tiredness Numeric Rating Scale (NRS)
Description: A participant-administered, single-item, 11-point horizontal scale anchored at 0 and 10, with 0 representing (no tiredness) and 10 representing (as bad as you can imagine). Participants rate their tiredness by selecting the one number that describes their worst level of tiredness during the past 24 hours. Total scores ranged from 0-10.
Time Frame: Baseline, Week 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 172 | 172 | 175
Units on a Scale | -1.1 (2.3) | -1.8 (2.7) | -2.0 (2.6)
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; Test type: Superiority or Other; p = 0.001, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05
Statistical Analysis 2: Comparison: Placebo vs Baricitinib 2 mg; Test type: Superiority or Other; p = 0.018, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05

18. Secondary Outcome: Change From Baseline in Worst Joint Pain NRS
Description: Participant-administered, single-item, 11-point horizontal scale anchored at 0 and 10, with 0 representing (no joint pain) and 10 representing (pain as bad as you can imagine). Participants rate their joint pain by selecting the one number that describes their worst level of joint pain during the past 24 hours. Total scores ranged from 0-10.
Time Frame: Baseline, Week 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 172 | 172 | 175
Units on a Scale | -1.2 (2.4) | -2.1 (2.5) | -2.5 (2.7)
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; Test type: Superiority or Other; p = 0.001, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05
Statistical Analysis 2: Comparison: Placebo vs Baricitinib 2 mg; Test type: Superiority or Other; p = 0.001, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05

19. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue Scale Scores
Description: The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scale is a brief 13-item, symptom-specific questionnaire that specifically assesses the participant's self-reported severity of fatigue and its impact upon daily activities and functioning. The FACIT-F uses a numeric rating scale of 0 (Not at all) to 4 (Very much) for each item to assess fatigue and its impact in the past 7 days. Total scores range from 0 to 52, with higher scores indicating less fatigue.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 170 | 170 | 174
Units on a Scale
  Week 12 | 5.9 (10.5) | 8.8 (10.0) | 8.5 (9.9)
  Week 24 | 6.6 (10.7) | 8.8 (10.4) | 9.7 (10.7)
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; Week 12; Test type: Superiority or Other; p = 0.005, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05
Statistical Analysis 2: Comparison: Placebo vs Baricitinib 2 mg; Week 12; Test type: Superiority or Other; p = 0.004, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05
Statistical Analysis 3: Comparison: Placebo vs Baricitinib 4 mg; Week 24; Test type: Superiority or Other; p = 0.002, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05
Statistical Analysis 4: Comparison: Placebo vs Baricitinib 2 mg; Week 24; Test type: Superiority or Other; p = 0.026, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05

20. Secondary Outcome: Change From Baseline in Mental Component Score (MCS), Physical Component Score (PCS) of the Medical Outcomes Study 36-Item Short Form Health Survey Version 2 Acute (SF-36v2 Acute)
Description: The SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, and 2 component scores (mental [MCS] and physical [PCS]). MCS consisted of social functioning, vitality, mental health, and role-emotional scales. PCS consisted of physical functioning, bodily pain, role-physical, and general health scales. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with higher scores indicating better health status.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 168 | 168 | 174
Units on a Scale
  Week 12 MCS | 1.6 (10.7) | 3.4 (9.7) | 2.4 (10.0)
  Week 24 MCS | 2.5 (10.8) | 3.2 (11.5) | 3.3 (10.6)
  Week 12 PCS | 3.3 (8.0) | 6.3 (8.8) | 6.4 (8.8)
  Week 24 PCS | 2.4 (8.2) | 6.4 (8.9) | 7.0 (9.3)
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; MCS Week 12; Test type: Superiority or Other; p = 0.448, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Baricitinib 2 mg; MCS Week 12; Test type: Superiority or Other; p = 0.058, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Baricitinib 4 mg; MCS Week 24; Test type: Superiority or Other; p = 0.446, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs Baricitinib 2 mg; MCS Week 24; Test type: Superiority or Other; p = 0.401, ANCOVA
Statistical Analysis 5: Comparison: Placebo vs Baricitinib 4 mg; PCS Week 12; Test type: Superiority or Other; p = 0.001, ANCOVA
Statistical Analysis 6: Comparison: Placebo vs Baricitinib 2 mg; PCS Week 12; Test type: Superiority or Other; p = 0.001, ANCOVA
Statistical Analysis 7: Comparison: Placebo vs Baricitinib 4 mg; PCS Week 24; Test type: Superiority or Other; p = 0.001, ANCOVA
Statistical Analysis 8: Comparison: Placebo vs Baricitinib 2 mg; PCS Week 24; Test type: Superiority or Other; p = 0.001, ANCOVA

21. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions-5 Level Scores
Description: European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) is a standardized measure of health status of the participant. The first component is a descriptive system of the respondent's health comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using the United Kingdom (UK) algorithm, with scores ranging from -0.594 to 1, and the United States (US) algorithm, with scores ranging from -0.109 to 1. A higher score indicates better health state. The second component is a self-perceived health score which is assessed using a VAS that ranged from 0 to 100 millimeter (mm), where 0 mm indicated the worst health you can imagine and 100 mm indicated the best health you can imagine.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 168 | 168 | 173
Units on a Scale
  Index Score (US Algorithm) Wk 12 (N=168,168,173) | 0.035 (0.167) | 0.080 (0.152) | 0.128 (0.148)
  Index Score (US Algorithm) Wk 24 (N=167,168,173) | 0.042 (0.166) | 0.082 (0.170) | 0.128 (0.157)
  Index Score (UK Algorithm) Wk 12 (N=168,168,173) | 0.052 (0.250) | 0.116 (0.224) | 0.191 (0.224)
  Index Score (UK Algorithm) Wk 24 (N=167,168,173) | 0.064 (0.245) | 0.122 (0.250) | 0.192 (0.237)
  Self-Perceived Health Wk 12 (N=168,168,173) | 4.1 (29.0) | 14.1 (24.2) | 10.3 (27.3)
  Self-Perceived Health Wk 24 (N=167,168,173) | 3.8 (27.8) | 11.4 (26.5) | 13.3 (29.0)
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; Week 12, US Algorithm; Test type: Superiority or Other; p = 0.001, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05
Statistical Analysis 2: Comparison: Placebo vs Baricitinib 2 mg; Week 12, US Algorithm; Test type: Superiority or Other; p = 0.001, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05
Statistical Analysis 3: Comparison: Placebo vs Baricitinib 4 mg; Week 24, US Algorithm; Test type: Superiority or Other; p = 0.001, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05
Statistical Analysis 4: Comparison: Placebo vs Baricitinib 2 mg; Week 24, US Algorithm; Test type: Superiority or Other; p = 0.003, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05
Statistical Analysis 5: Comparison: Placebo vs Baricitinib 4 mg; Week 12, UK Algorithm; Test type: Superiority or Other; p = 0.001, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05
Statistical Analysis 6: Comparison: Placebo vs Baricitinib 2 mg; Week 12, UK Algorithm; Test type: Superiority or Other; p = 0.001, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05
Statistical Analysis 7: Comparison: Placebo vs Baricitinib 4 mg; Week 24, UK Algorithm; Test type: Superiority or Other; p = 0.001, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05
Statistical Analysis 8: Comparison: Placebo vs Baricitinib 2 mg; Week 24, UK Algorithm; Test type: Superiority or Other; p = 0.002, ANCOVA — a priori p-value significance threshold: 2-sided ≤0.05

22. Secondary Outcome: Percentage Change From Baseline in Work Productivity and Activity Impairment-Rheumatoid Arthritis (WPAI-RA) Scores
Description: The WPAI-RA participant questionnaire was developed to measure the effect of general health and symptom severity on work productivity and regular activities in the 7 days prior to the visit. Using 6 questions, it yields four types of scores: absenteeism (work time missed), presenteeism (impairment at work), work productivity loss (overall work impairment), and activity impairment, with outcomes expressed as impairment percentages. Percentage work time missed absenteeism: Q2/(Q2+Q4)*100, Percentage impairment while working presenteeism: Q5/10*100; Percentage overall work impairment work productivity loss: Q2/(Q2+Q4)+[(1-Q2/(Q2+Q4))x(Q5/10)]*100; Percentage activity impairment activity impairment: Q6/10*100. Higher numbers indicate greater impairment and less productivity, that is, worse outcomes.
Time Frame: Baseline, Week 12, Week 24
Population: mITT population includes all randomized participants who received at least 1 dose of the study drug. Participants were analyzed according to the study drug to which they were randomized.
Measure: Mean (Standard Deviation); unit: Percentage of Impairment
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 176 | 174 | 177
Percentage of Impairment
  Absenteeism Week 12 | 3.2 (23.8) | -6.7 (26.6) | -6.5 (22.1)
  Absenteeism Week 24 | 0.9 (12.4) | -1.9 (31.4) | -2.3 (29.5)
  Presenteeism Week 12 | -4.1 (26.4) | -12.0 (24.0) | -10.5 (24.0)
  Presenteeism Week 24 | -7.1 (30.5) | -11.4 (24.9) | -15.6 (25.4)
  Work Productivity Loss Week 12 | -4.2 (27.8) | -13.7 (26.7) | -12.3 (24.8)
  Work Productivity Loss Week 24 | -6.0 (33.4) | -13.2 (27.6) | -14.8 (32.4)
  Activity Impairment Week 12 | -10.4 (22.8) | -16.0 (25.5) | -18.1 (24.8)
  Activity Impairment Week 24 | -15.7 (25.5) | -20.8 (23.7) | -25.8 (25.2)
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; Absenteeism Week 12; Test type: Superiority or Other; p = 0.362, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Baricitinib 2 mg; Absenteeism Week 12; Test type: Superiority or Other; p = 0.170, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Baricitinib 4 mg; Absenteeism Week 24; Test type: Superiority or Other; p = 0.753, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs Baricitinib 2 mg; Absenteeism Week 24; Test type: Superiority or Other; p = 0.715, ANCOVA
Statistical Analysis 5: Comparison: Placebo vs Baricitinib 4 mg; Presenteeism Week 12; Test type: Superiority or Other; p = 0.077, ANCOVA
Statistical Analysis 6: Comparison: Placebo vs Baricitinib 2 mg; Presenteeism Week 12; Test type: Superiority or Other; p = 0.058, ANCOVA
Statistical Analysis 7: Comparison: Placebo vs Baricitinib 4 mg; Presenteeism Week 24; Test type: Superiority or Other; p = 0.232, ANCOVA
Statistical Analysis 8: Comparison: Placebo vs Baricitinib 2 mg; Presenteeism Week 24; Test type: Superiority or Other; p = 0.534, ANCOVA
Statistical Analysis 9: Comparison: Placebo vs Baricitinib 4 mg; Work Productivity Loss Week 12; Test type: Superiority or Other; p = 0.079, ANCOVA
Statistical Analysis 10: Comparison: Placebo vs Baricitinib 2 mg; Work Productivity Loss Week 12; Test type: Superiority or Other; p = 0.070, ANCOVA
Statistical Analysis 11: Comparison: Placebo vs Baricitinib 4 mg; Work Productivity Loss Week 24; Test type: Superiority or Other; p = 0.327, ANCOVA
Statistical Analysis 12: Comparison: Placebo vs Baricitinib 2 mg; Work Productivity Loss Week 24; Test type: Superiority or Other; p = 0.479, ANCOVA
Statistical Analysis 13: Comparison: Placebo vs Baricitinib 4 mg; Activity Impairment Week 12; Test type: Superiority or Other; p = 0.001, ANCOVA
Statistical Analysis 14: Comparison: Placebo vs Baricitinib 2 mg; Activity Impairment Week 12; Test type: Superiority or Other; p = 0.005, ANCOVA
Statistical Analysis 15: Comparison: Placebo vs Baricitinib 4 mg; Activity Impairment Week 24; Test type: Superiority or Other; p = 0.001, ANCOVA
Statistical Analysis 16: Comparison: Placebo vs Baricitinib 2 mg; Activity Impairment Week 24; Test type: Superiority or Other; p = 0.030, ANCOVA

23. Secondary Outcome: Population Pharmacokinetics (PK): Maximum Concentration at Steady State of Dosing (Cmax,ss) of Baricitinib
Time Frame: Week 0 (Baseline): 15 min. post-dose, 1 hour post-dose. Week 4 (Day 28 ±2 days): 2 to 4 hours post-dose. Week 8 (Day 56 ±3 days): 4 to 6 hours post-dose. Week 12 (Day 84 ±3 days): Pre-dose. Week 24 (Day 168 ±5 days): Pre-dose.
Population: All randomized participants who received at least 1 dose of study drug (during study or rescue treatment) with evaluable PK data. Participants who initially received 2 mg with renal impairment were randomized to 4mg (N=11). Participants starting on 4mg (N=177) and participants rescued to 4mg (N=33) are included in the PK baricitinib 4 mg arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles/Liter (nmol/L)
Groups:
- Baricitinib 2 mg: Baricitinib 2 mg administered PO QD through Week 24 (N=185). Participants who were randomized to 4mg (N=11) but actually received 2 mg due to moderate renal impairment were included in the 2-mg group.
  Participants continued to take background cDMARD therapy throughout study.
- Baricitinib 4 mg: Baricitinib 4 mg administered PO QD through Week 24 (n=177). Participants rescued to 4mg (N=33) are included in the PK baricitinib 4 mg arm.
  Participants continued to take background cDMARD therapy throughout study.
Arm/Group | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 185 | 210
nanomoles/Liter (nmol/L) | 65.6 (21.4) | 130 (19.3)

24. Secondary Outcome: Population PK: Area Under the Concentration Curve Versus Time at a Dosing Interval at Steady State (AUCtau,ss) of Baricitinib
Time Frame: as for outcome 23
Population: All randomized participants who received at least 1 dose of study drug (during study or rescue treatment) with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles*hour/Liter (nmol*h/L)
Arm/Group | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 185 | 210
nanomoles*hour/Liter (nmol*h/L) | 615 (43.1) | 1140 (38.7)

ADVERSE EVENTS:
Groups:
- Placebo -Treatment Period: Placebo administered PO QD through Week 24. Participants continued to take background cDMARD therapy throughout study.
- Baricitinib 2 mg - Treatment Period: Baricitinib 2mg administered PO QD through Week 24. Participants continued to take background cDMARD therapy throughout study.
- Baricitinib 4 mg - Treatment Period; Rescue Period: Baricitinib 4 mg administered PO QD through Week 24. Participants continued to take background cDMARD therapy throughout study.
- Placebo - Follow Up Period; Baricitinib 2 mg - Follow Up Period; Baricitinib 4 mg - Follow Up Period: No study drug received. Participants return for safety follow-up visit 28 days after the last dose of study drug.
Arm/Group | Placebo -Treatment Period | Baricitinib 2 mg - Treatment Period | Baricitinib 4 mg - Treatment Period | Rescue Period | Placebo - Follow Up Period | Baricitinib 2 mg - Follow Up Period | Baricitinib 4 mg - Follow Up Period
Serious Adverse Events (participants affected / at risk) | 14/176 | 8/174 | 19/177 | 2/127 | 1/19 | 1/9 | 0/20
Other Adverse Events (participants affected / at risk) | 79/176 | 105/174 | 102/177 | 6/127 | 2/19 | 4/9 | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo -Treatment Period (N=176) | Baricitinib 2 mg - Treatment Period (N=174) | Baricitinib 4 mg - Treatment Period (N=177) | Rescue Period (N=127) | Placebo - Follow Up Period (N=19) | Baricitinib 2 mg - Follow Up Period (N=9) | Baricitinib 4 mg - Follow Up Period (N=20)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device complication (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulval abscess (Infections and infestations) | 0/145 (0) | 0/137 (0) | 1/149 (1) | 0/113 (0) | 0/16 (0) | 0 (0) | 0/18 (0)
Accident at work (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basilar artery thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient global amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebral artery thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo -Treatment Period (N=176) | Baricitinib 2 mg - Treatment Period (N=174) | Baricitinib 4 mg - Treatment Period (N=177) | Rescue Period (N=127) | Placebo - Follow Up Period (N=19) | Baricitinib 2 mg - Follow Up Period (N=9) | Baricitinib 4 mg - Follow Up Period (N=20)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Episcleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 7 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (5) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 10 (10) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 7 (9) | 10 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (5) | 6 (6) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 7 (8) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 6 (7) | 6 (7) | 10 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervicitis (Infections and infestations) | 0/145 (0) | 0/137 (0) | 0/149 (0) | 0/113 (0) | 0/16 (0) | 0 (0) | 1/18 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 4 (4) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 4 (4) | 8 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (7) | 12 (13) | 9 (10) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 8 (8) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 15 (17) | 9 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (6) | 7 (10) | 8 (10) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0/145 (0) | 3/137 (3) | 0/149 (0) | 0/113 (0) | 0/16 (0) | 0 (0) | 0/18 (0)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 4 (4) | 6 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 3 (4) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (8) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (6) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 7 (8) | 5 (6) | 8 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 11 (12) | 17 (17) | 12 (12) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (6) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 7 (7) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days